CLINICAL TRIAL: NCT02478515
Title: Evaluation of Visual Acuity Improvement of a PRN Regimen Using Ranibizumab for Macular Edema Due to Ischemic and Non- Ischemic Branch Retinal Vein Occlusion.
Brief Title: Evaluation of the Usefulness of a PRN Regimen Using Ranibizumab for Macular Edema Due to Branch Retinal Vein Occlusion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nagoya City University (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Yuichiro Ogura, Professor, Nagoya City University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRNNCU001
Record Dates: First submitted 2015-01-26; First posted 2015-06-23 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2016-10

CONDITIONS: Branch Retinal Vein Occlusion
Keywords: ranibizumab; PRN regimen; macular edema; branch retinal vein occlusion
MeSH Terms: conditions — Retinal Vein Occlusion; Macular Edema | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intraviteal Ranibizumab 0.5mg (Experimental): Intraviteal Ranibizumab 0.5mg
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — Intraviteal injection of 0.5mg ranibizumab
  Other Names: Lucentis

SUMMARY:
Monthly intravitreal ranibizumab (IVR) during the first 6 month had great effect for macular edema with branch retinal vein occlusion (BVO) both in visual and anatomical outcome. It is expected that similar results could be obtained by less frequent IVR. The purpose of this study is to investigate if IVR by PRN is as effective as by monthly. In addition, the investigators are going to study the relationship between macular edema and the size and location of retinal non-perfusion area.

DETAILED DESCRIPTION:
It was demonstrated in BRAVO study that IVR had great effect for macular edema with BVO both in visual and anatomical outcome. However IVR was done monthly for all patients (except Sham group) during the first 6 months in BRAVO study. It is expected that similar results could be obtained by less frequent IVR, and if so, it will contribute to reduce patient's burden and medical cost. Thus it is necessary to determine the optimal regimen of IVR therapy.

In this study, considering the medical and social circumstances in Japan, the investigators are going to investigate if IVR by PRN is as effective as BRAVO study.In addition, the investigators are going to study the relationship between macular edema and the size and location of retinal non-perfusion area (NPA), because VEGF is thought to be released from non-perfused retinal tissue, and VEGF production may be correlated with NPA size and location. The investigators are going to measure the size of NPA semi-quantatively by ultra wide field fluorescein angiography (UWFA) using Optos 200Tx. Then the relationship with macular edema will be studied. The effect of ranibizumab to NPA is controversial. In this study, it will be investigated, too.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Macula edema secondary to BRVO
* BCVA of 77 to 20 letters assessed with the use of ETDRS charts
* CRT ≧250μm

Exclusion Criteria:

* Previous treatment with anti-VEGF drugs or corticosteroid or grid laser photocoagulation (study eye)
* History of vitrectomy surgery, submacular surgery, or other surgical intervention for RVO
* Ocular disorders in the study eye that may confound interpretation of study results
* BCVA over 77 letters between screening and Day 0
* The pregnant or lactating woman

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-01; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Visual acuity | One years

SECONDARY OUTCOMES:
central foveal thickness | One and two years
Visual acuity | Two years

OTHER OUTCOMES:
size and location of retinal non-perfusion area | one and two years

CONTACTS AND LOCATIONS:
Overall Officials: Yuichiro Ogura, Study Chair — Nagoya City Univsersity
Locations (1):
- Nagoya City Univsersity, Nagoya, Aichi-ken, Japan

IPD SHARING:
Plan to Share IPD: No